CLINICAL TRIAL: NCT00006129
Title: Randomized Study of Testosterone and Progressive Resistance Exercise in Men With Burn Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/15290; UTMB-97-284; UTMB-GCRC-474
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Burns
Keywords: burns; dermatologic disorders; rare disease
MeSH Terms: conditions — Burns; Skin Diseases; Rare Diseases | interventions — Testosterone

INTERVENTIONS:
Drug: testosterone

SUMMARY:
OBJECTIVES: I. Determine whether testosterone normalization ameliorates muscle protein hypercatabolism by increasing net protein synthesis in men with burn injury.

II. Determine whether the effectiveness of testosterone is enhanced by stimulation of inward amino acid transport as a consequence of hyperaminoacidemia in these men.

III. Determine whether testosterone normalization during hospitalization minimizes the need for rehabilitation by increasing net protein synthesis and preserving skeletal muscle in these men.

IV. Determine whether testosterone normalization after hospital discharge and throughout convalescence increases muscle strength and lean body mass after burn injury by increasing net protein synthesis.

V. Determine whether testosterone combined with progressive resistance exercise during convalescence confers added benefits on muscle protein synthesis, and in turn, lean body mass and muscle strength in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are stratified according to percent of total body surface area (TBSA) burned (no more than 40% vs more than 40%).

Patients receive standard inpatient burn care. During hospitalization, patients are randomized to one of two treatment arms:

Arm I: Patients receive testosterone intramuscularly (IM) weekly for 2-3 weeks during hospitalization.

Arm II: Patients receive standard care only during hospitalization.

After hospital discharge, patients with burns covering no more than 40% of TBSA are randomized to arm III, IV, or V, whereas patients with burns covering more than 40% of TBSA are randomized to arm III or V.

Arm III: Patients receive testosterone IM every 2 weeks for 2 months.

Arm IV: Patients receive testosterone as in arm III. Patients perform progressive resistance (weight lifting) exercises 3 times a week for 2 months concurrently with testosterone therapy.

Arm V.: Patients receive standard convalescence care only.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Second degree or worse burn injury Percent of total body surface area burned and degree of burn(s) must be carefully quantified

--Patient Characteristics--

Cardiovascular: No limiting or unstable angina No myocardial infarction within the past 6 months No horizontal or downsloping ST segment depression greater than 0.2 mV and/or frequent or repetitive arrhythmias (defined as more than 10 premature ventricular contractions per minute) No hypertension that is uncontrolled by one blood pressure medication No prior arrhythmia or valvular disease requiring treatment

Other: No history of prostate cancer or indication of an occult carcinoma, defined by PSA greater than 4.0 micrograms/L

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Arny A. Ferrando, Study Chair — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States